CLINICAL TRIAL: NCT00243347
Title: An Exploratory, Open-Lael Study to Assess the Effects of AZD2171 on Tumors and Biomarkers in Patients With Previously Untreated or Recurrent Non-small Cell Lung Cancer (NSCLC) or Patients With Metastatic or Recurrent Head and Neck Cancer (HNC)
Brief Title: The Effects of AZD2171 in Patients With Non-Small Cell Lung Cancer or Head & Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00015
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-08

CONDITIONS: Carcinoma; Non-Small-Cell Lung Carcinoma; Head and Neck Neoplasms
Keywords: RECENTIN
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — cediranib

INTERVENTIONS:
Drug: AZD2171 — oral tablet
  Other Names: cediranib; RECENTIN™

SUMMARY:
This study is to examine the effects on tumors of AZD2171, in the treatment of NSCLC or HNC. The safety and tolerability of AZD2171 will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed head and neck cancer (HNC) or unresectable stage IIIb or IV non-small cell lung cancer (NSCLC)
* At least one lesion able to be used for tumor biopsy and to be measured by FDG-PET Scan
* Considered suitable for treatment of NSCLC with no prior biological or immunological therapy for disease
* Or considered suitable for treatment for metastatic or recurrent HNC with no prior biological or immunological therapy for disease

Exclusion Criteria:

* NSCLC: Have received more than 2 previous chemotherapy regimens or have received the last chemotherapy or radiotherapy within 28 days of first dose of AZD2171
* HNC: Previous chemotherapy or radiotherapy if received 28 days of first dose of AZD2171
* Untreatable, unstable brain or meningeal metastases.
* Abnormal liver and kidney blood chemistries
* History of poorly controlled hypertension with resting blood pressure of >150/100
* Recent (< 14 days) major surgery or a surgical incision not fully healed
* Diabetes patients with type I insulin dependent diabetes or poorly controlled type II
* Significant hemorrhage or hemoptysis
* Presence of necrotic/hemorrhagic tumor or metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (2):
- Research Site, Houston, Texas, United States
- Research Site, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Cediranib 30 mg: Cediranib 30mg/Day
Period: Overall Study
Arm/Group | Cediranib 30 mg
Started | 19 (Treated)
Completed | 0 (Completed study)
Not Completed | 19
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 5
Not completed — Condition worsened | 7

BASELINE CHARACTERISTICS:
Arm/Group | Cediranib 30 mg
Number analyzed (Participants) | 19
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Standardised Uptake Value (SUVmax) as Measured by 2-[F-18]-Fluoro-2-deoxy-D-glucose Positron Emission Tomography (FDG-PET)
Description: Percentage Change from baseline in Standardised Uptake Value (SUVmax) at Day 22, as Measured by 2-[F-18]-fluoro-2-deoxy-D-glucose positron emission tomography (FDG-PET) Response ((Day 22 SUVmax value - baseline SUVmax value)/baseline SUVmax value)*100
Time Frame: Randomisation until Day 22
Population: Of the 19 patients, only 17 patients were evaluable for FDG-PET analysis. To be evaluable for FDG-PET, patients had to have FDG-PET data collected at Day 1 and at least one post-baseline visit.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage change in SUVmax
Arm/Group | Cediranib 30 mg
Number analyzed (Participants) | 17
Percentage change in SUVmax | -18.386 [-35.496 to 3.263]

2. Secondary Outcome: Change From Baseline in Mean Arterial Blood Pressure (MAP)
Description: Change from baseline in mean arterial blood pressure (MAP) (MAP value at Day 22 - MAP value at baseline).
Time Frame: Randomisation until Day 22
Population: Of the 19 patients, only 17 patients were evaluable MAP analysis. To be evaluable for MAP analysis, patients had to have MAP data collected at Day 1 and at least one post-baseline visit.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Cediranib 30 mg
Number analyzed (Participants) | 17
mmHg | 6.853 (1.010) [1.010 to 12.696]

ADVERSE EVENTS:
Arm/Group | Cediranib 30 mg
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30 mg (N=19)
Anaemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tongue Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Acquired Tracheo-Oesophageal Fistula (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30 mg (N=19)
Lymphopenia (Blood and lymphatic system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Enteritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Asthenia (General disorders) | 4
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 1
Localised Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Oral Candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Blood Corticotrophin Increased (Injury, poisoning and procedural complications) | 4
Weight Decreased (Injury, poisoning and procedural complications) | 4
Blood Thyroid Stimulating Hormone Increased (Injury, poisoning and procedural complications) | 2
Blood Thyroid Stimulating Hormone Decreased (Injury, poisoning and procedural complications) | 1
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 1
Urine Colour Abnormal (Injury, poisoning and procedural complications) | 1
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Aphonia (Nervous system disorders) | 1
Cervical Root Pain (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 8
Ketonuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Skin Reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.